CLINICAL TRIAL: NCT01029366
Title: Pilot Study of Redirected Autologous T-cells Engineered to Contain Anti-CD19 Attached to TCR and 4-1BB Signaling Domains in Patient With Chemotherapy Resistant or Refractory CD19+ Leukemia and Lymphoma
Brief Title: CART19 to Treat B-Cell Leukemia or Lymphoma That Are Resistant or Refractory to Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC04409, 809517; NCI-2009-01357; NCT00891215 (obsolete NCT alias)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2019-06

CONDITIONS: Hematopoietic/Lymphoid Cancer; Adult Acute Lymphoblastic Leukemia in Remission; B-cell Adult Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CART-19 CLL (Experimental): CART-19 (autologous T cells transduced with CD19 TCR-ζ/4-1BB vector) administered as an IV infusion days 0, 1, 2 and 11 in the absence of disease progression or unacceptable toxicity.Minimum/maximum total dose: 1.5x10^7 / 5x10^9 administered to patients with chronic Lymphocytic Leukemia (CLL) and Acute Lymphoblastic Leukemia (ALL).
  Interventions: Biological: CART-19
- CART-19 ALL (Experimental): CART-19 (autologous T cells transduced with CD19 TCR-ζ/4-1BB vector) administered as an IV infusion days 0, 1, 2 and 11 in the absence of disease progression or unacceptable toxicity.Minimum/maximum total dose: 1.5x10^7 / 5x10^9 administered to patients with chronic Lymphocytic Leukemia (CLL) and Acute Lymphoblastic Leukemia (ALL).
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — Autologous T cells purified from the peripheral blood mononuclear cells of subjects, transduced with TCR-ζ/4-1BB lentiviral vector, expanded in vitro and then frozen for future administration.

SUMMARY:
This is a Pilot/Phase I, single arm, single center, open label study to determine the safety, efficacy and cellular kinetics of CART19 (CTL019) in chemotherapy resistant or refractory CD19+ leukemia and lymphoma subjects. The study consists of three Phases:

1) a Screening Phase, followed by 2) an Intervention/Treatment Phase consisting of apheresis, lymphodepleting chemotherapy (determined by the Investigator and based on subject's disease burden and histology, as well as on the prior chemotherapy history received), infusions of CTL019, tumor collection by bone marrow aspiration or lymph node biopsy (optional, depending on availability), and 3) a Follow-up Phase.

The suitability of subjects' T cells for CTL019 manufacturing was determined at study entry.

Subjects with adequate T cells were leukapheresed to obtain large numbers of peripheral blood mononuclear cells for CTL019 manufacturing. The T cells were purified from the peripheral blood mononuclear cells, transduced with TCR-ζ/4-1BB lentiviral vector, expanded in vitro and then frozen for future administration. The number of subjects who had inadequate T cell collections, expansion or manufacturing compared to the number of subjects who had T cells successfully manufactured is a primary measure of feasibility of this study.

Unless contraindicated and medically not advisable based on previous chemotherapy, subjects were given conditioning chemotherapy prior to CTL019 infusion. The chemotherapy was completed 1 to 4 days before the planned infusion of the first dose of CTL019.

Up to 20 evaluable subjects with CD19+ leukemia or lymphoma were planned to be dosed with CTL019. A single dose of CTL019 (consisting of approximately 5x10^9 total cells, with a minimal acceptable dose for infusion of 1.5x10^7 CTL019 cells) was to be given to subjects as fractions (10%, 30% and 60% of the total dose) on Day 0, 1 and 2. A second 100% dose of CTL019 was initially permitted to be given on Day 11 to 14 to subjects, providing they had adequate tolerance to the first dose and sufficient CTL019 was manufactured.

DETAILED DESCRIPTION:
Primary objectives:

1. To evaluate the safety and feasibility of a single target dose of 5 times 10e9 total cells, acceptable range of 1.5 times 10e7 to 5 times 10e9 total cells comprised of autologous CART-19 cells that express the TCR zeta and 4-1 BB costimulatory domain.

Secondary objectives:

1. Proof of mechanism: determine if 2nd generation CAR expressing 4-1BB costimulation domains have improved persistence in patients.
2. Proof of concept: determine the effects of CART-19 on CD19 expression in vivo.
3. Proof of bioactivity: Evaluate changes in systemic soluble immune factors in patients
4. Proof of bioactivity: Evaluate impact of CART19 treatment on tumor burden
5. Explore whether CART-19 cells retain anti-tumor activity in vivo.
6. Determine if host immunity develops against CART-19.
7. Characterize the relative subsets of CART-19 T cells (Tcm, Tem, and Treg).
8. Describe survival and response rates

ELIGIBILITY:
Inclusion

* Male and female subjects with CD19+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled
* CD19+ leukemia or lymphoma
* ALL in CR2 or CR3 and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor
* Follicular lymphoma, previously identified as CD19+:
* At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy
* Stage III-IV disease
* Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year)
* Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc)
* CLL:
* At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy. Patients with high risk disease manifested by deletion chromosome 17p will be eligible if they fail to achieve a CR to initial therapy or progress within 2 years of 1 prior
* Less than 2 years between last chemotherapy and progression (i.e. most recent progression free interval < 2 years)
* Not eligible or appropriate for conventional allogeneic SCT
* Patients who achieve only a partial response to FCR as initial therapy will be eligible.
* Mantle cell lymphoma:
* Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
* Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc...)
* Relapsed after prior autologous SCT
* B-cell prolymphocytic leukemia (PLL) with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT
* Diffuse large cell lymphoma, previously identified as CD19+:
* Residual disease after primary therapy and not eligible for autologous SCT
* Relapsed after prior autologous SCT
* Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate of conventional allogeneic or autologous SCT
* Expected survival > 12 weeks
* Creatinine < 2.5 mg/dl
* ALT/AST < 3x normal
* Bilirubin < 2.0 mg/dl
* Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion

* Pregnant or lactating women
* The safety of this therapy on unborn children is not known
* Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD28 costimulation
* Any uncontrolled active medical disorder that would preclude participation as outlined
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03-17 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Frey NV, Shaw PA, Hexner EO, Pequignot E, Gill S, Luger SM, Mangan JK, Loren AW, Perl AE, Maude SL, Grupp SA, Shah NN, Gilmore J, Lacey SF, Melenhorst JJ, Levine BL, June CH, Porter DL. Optimizing Chimeric Antigen Receptor T-Cell Therapy for Adults With Acute Lymphoblastic Leukemia. J Clin Oncol. 2020 Feb 10;38(5):415-422. doi: 10.1200/JCO.19.01892. Epub 2019 Dec 9. PMID 31815579
- [Derived] van Bruggen JAC, Martens AWJ, Fraietta JA, Hofland T, Tonino SH, Eldering E, Levin MD, Siska PJ, Endstra S, Rathmell JC, June CH, Porter DL, Melenhorst JJ, Kater AP, van der Windt GJW. Chronic lymphocytic leukemia cells impair mitochondrial fitness in CD8+ T cells and impede CAR T-cell efficacy. Blood. 2019 Jul 4;134(1):44-58. doi: 10.1182/blood.2018885863. Epub 2019 May 10. PMID 31076448
- [Derived] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start/End Dates 17-Mar-2010 to 06-Jul-2015
Groups:
- Chronic Lymphocytic Leukemia (CLL) Subjects; Acute Lymphocytic Leukemia (ALL) Subjects: Patients receive CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:41BB administered on days 0, 1, 2 and 11 in the absence of disease progression or unacceptable toxicity laboratory biomarker analysis polymerase chain reaction reverse transcriptase-polymerase chain reaction anti-CD19-CAR retroviral vector-transduced autologous T cells: Given IV genetically engineered lymphocyte therapy. Subjects were given minimum/maximum total dose: 1.5x10⁷/ 5x10⁹.
Period: Overall Study
Arm/Group | Chronic Lymphocytic Leukemia (CLL) Subjects | Acute Lymphocytic Leukemia (ALL) Subjects
Started | 18 | 8
Completed | 14 | 6
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 1
Not completed — disease progression | 2 | 0
Not completed — manufacturing failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CLL Subjects; ALL Subjects: Patients receive CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:41BB administered on days 0, 1, 2 and 11 in the absence of disease progression or unacceptable toxicity laboratory biomarker analysis polymerase chain reaction reverse transcriptase-polymerase chain reaction anti-CD19-CAR retroviral vector-transduced autologous T cells: Given IV genetically engineered lymphocyte therapy
- Total: Total of all reporting groups
Arm/Group | CLL Subjects | ALL Subjects | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 7 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 12 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 14 | 4 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 5 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 5 years
Measure: Number; unit: participants
Groups:
- All Participants: Patients receive CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:41BB administered on days 0, 1, 2 and 11 in the absence of disease progression or unacceptable toxicity laboratory biomarker analysis
  polymerase chain reaction
  reverse transcriptase-polymerase chain reaction
  anti-CD19-CAR retroviral vector-transduced autologous T cells: Given IV
  genetically engineered lymphocyte therapy
Arm/Group | All Participants
Number analyzed (Participants) | 20
participants | 20

2. Secondary Outcome: Overall Response Summary
Description: Efficacy assessments for ALL were performed based on bone marrow and blood morphologic criteria and physical examination findings. The definitions for response are primarily based on the standardized response criteria defined by National Comprehensive Cancer Network (NCCN) Guidelines (NCCN, 2013 v.1).
  Efficacy assessments for CLL were based on lymphadenopathy, hepatomegaly, splenomegaly, bone marrow and blood morphologic and laboratory assessments. The response criteria are consistent with NCCN Guidelines Version 2.2012 CLL/SLL, which is based on the 2008 International Workshop Group on CLL (IWCLL) revisions of the original guidelines for evaluating disease response released in 1996 by the National Cancer Institute Working Group (NCI/WG).
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | CLL Subjects | ALL Subjects
Number analyzed (Participants) | 14 | 6
percentage of participants
  Complete Remission | 21.4 | 83.4
  Partial Remission | 21.4 | 0
  No Remission | 57.1 | 16.7
  Overall Response Rate | 42.9 | 83.3

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events during post-infusion period, regardless of study drug relationship, by primary system organ class and maximum CTC grade
Groups:
- Chronic Lymphocytic Leukemia; Acute Lymphocytic Leukemia: CART-19 (autologous T cells transduced with CD19 TCR-ζ/4-1BB vector) administered as an IV infusion. Minimum/maximum total dose: 1.5x10^7 / 5x10^9.
Arm/Group | Chronic Lymphocytic Leukemia | Acute Lymphocytic Leukemia
Serious Adverse Events (participants affected / at risk) | 14/14 | 6/6
Other Adverse Events (participants affected / at risk) | 14/14 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia (N=14) | Acute Lymphocytic Leukemia (N=6)
Cytokine Release Syndrome (Immune system disorders) | 6 (6) | 5 (5) — Grading of this event was performed using a modified grading scale based upon CRS in the context of the experimental agent.
pyrexia (General disorders) | 4 (4) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Clostridium difficle infection (Infections and infestations) | 1 (1) | 0 (0)
Confusion State (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Histocytosis Haematophagic (Investigations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Influenza like illness (Infections and infestations) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomas Infection (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia (N=14) | Acute Lymphocytic Leukemia (N=6)
Fatigue (General disorders) | 13 (13) | 2 (2)
Pyrexia (General disorders) | 11 (11) | 2 (2)
Blood Albumin decreased (Investigations) | 8 (8) | 1 (1)
Chills (General disorders) | 8 (8) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 8 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 8 (8) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 8 (8) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Odema Peripheral (General disorders) | 7 (7) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Blood Calcium decreased (Investigations) | 6 (6) | 1 (1)
Blood Sosoim decreased (Investigations) | 6 (6) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood Glucose increased (Investigations) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Blood Glucose decreased (Investigations) | 4 (4) | 0 (0)
Blood Magnesium decreased (Investigations) | 4 (4) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (2)
hypertension (Vascular disorders) | 4 (4) | 0 (0)
Hypomagnesaemia (Investigations) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
ATrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Blood Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0)
blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0)
Blood phosphorous decreased (Investigations) | 3 (3) | 3 (3)
Blood urinc acid increased (Investigations) | 3 (3) | 0 (0)
Confusion state (Psychiatric disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
platelet count decreased (Investigations) | 3 (3) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes